CLINICAL TRIAL: NCT05253742
Title: Fetal MRI Acquisition and Sequence Development
Acronym: FMASD
Status: Not yet recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Andre van der Kouwe, PhD, Dr. Andre van der Kouwe, Massachusetts General Hospital
Other Study IDs: 2021P001433
Record Dates: First submitted 2022-01-11; First posted 2022-02-24 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Pregnancy Related
Keywords: MRI; Fetus; Uterus; Placenta; Brain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women presenting for MRI: Alternative motion-robust MR imaging sequences and procedures for automatic positioning while be tested during fetal brain imaging
  Interventions: Other: No intervention - the investigators are evaluating a new image acquisition method on an MRI scanner

INTERVENTIONS:
Other: No intervention - the investigators are evaluating a new image acquisition method on an MRI scanner — The investigators will evaluate the performance of a modified MRI acquisition method against an existing method in fetal imaging in volunteers

SUMMARY:
Testing of new magnetic resonance imaging (MRI) pulse sequences (image acquisition software) for imaging the fetus to improve workflow and image quality in fetal imaging and diagnosis. The investigators would like to develop novel MRI approaches to enhance fetal imaging with MRI, in the presence of motion. As part of technical development, the investigators plan to develop methods to improve structural T1 and T2 weighted images, MR angiography, diffusion and spectroscopy measurements of the fetus.

DETAILED DESCRIPTION:
Fetal MRI has become a critical tool for both studying the early development of the human brain and resolving diagnostic ambiguities that may remain after routine ultrasound exams. Due to its excellent soft-tissue contrast and the absence of harmful ionizing radiation, MRI is preferable to computed tomography for neuroimaging. Unfortunately, fetal and maternal motion limit fetal MRI to rapid two-dimensional (2D) sequences with thick slices such as half-Fourier single-shot turbo spin echo (HASTE). Although these sequences decrease the impact of motion during the sub-second acquisition of individual slices, multiple slices are needed, and contiguous orthogonal scans are challenging as motion occurs between slices. Typically, >38% of acquisitions are discarded because of corrupted geometry and artifacts.

In this project the investigators will develop software that runs on the Siemens MRI scanner. This software will improve the workflow for fetal imaging i.e. for imaging the fetus in utero. Fetal imaging in its current form is inefficient due to the frequent motion of the fetus during the imaging procedure. In this project the investigators will develop automated methods for alignment and tracking of the fetus during imaging, to more efficiently image the fetus and to obtain better image quality in a shorter examination. The investigators are specifically interested in the fetal brain, but these methods may be generalized to all fetal organ systems. The investigators will install the software on the scanner and test these methods with volunteers.

ELIGIBILITY:
Eligibility will be determined prior to the scan session by a pre-screening interview conducted either via telephone or in person asking about MR contraindications.

Participants will be excluded from study entry or study completion when any of the following exclusion criteria are met at any time of screening or enrollment:

* Claustrophobia sufficient to interfere with MRI or render the subject unable to complete an MRI scan
* MRI contraindications (e.g., magnetically or mechanically activated implants)
* Weight greater than or equal to 300lbs (weight limit of the MRI table)
* Non-English speaking
* Neurological conditions (i.e. epilepsy, multiple sclerosis, neurodegenerative diseases, memory disorders, brain tumor)
* Past incidence of stroke or heart attack
* Severe hypertension, blood disorders, advanced diabetes mellitus, or advanced cardiovascular disease
* Hospitalization within 6 weeks prior to enrollment
* Significant acute and/or chronic medical conditions, current use of medications that indicate the existence of significant medical conditions, and other unspecified reasons that make the subject unsuitable for enrollment at the discretion at the PI and a consulting MD.

Pregnant mothers with the following features will be excluded.

* Mothers with contraindication to MRI (such as pacemaker, metal in body, exceeding scanner weight or bore diameter limits (550lbs, 70cm))
* Mothers with claustrophobia
* Mothers medically unstable for the MRI study

Ages: 13 Weeks to 40 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Pregnant women presenting for imaging of the fetus
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-05-31 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Image alignment in fetal MRI | Five year K99/R00 project
  Evaluation of image alignment with automatical positioning in MRI
Tracking quality in fetal MRI | Five year K99/R00 project
  Evaluation of image quality with motion tracking in MRI

IPD SHARING:
Plan to Share IPD: No
The investigators will share data if requested as permitted by the Massachusetts General Brigham (MGB) Institutional Review Board (IRB).